CLINICAL TRIAL: NCT04296318
Title: Protocol for COPE-WEL Observational Validation Trial COPD Exacerbation Alert System With urinE anaLysis - Clinical Validation of the Headstart® Test System for Early Detection of Exacerbations in Moderate/Severe COPD Patients
Brief Title: COPD Exacerbation Alert System With urinE anaLysis Using the HEADSTART Device
Acronym: COPE-WEL
Status: Terminated | Type: Observational
Why Stopped: Business decision
Sponsor: Mologic Ltd (Industry)
Collaborators: University Hospitals, Leicester (Other)
Responsible Party: Sponsor
Other Study IDs: Headstart COPE-WEL MSR030/046
Record Dates: First submitted 2020-03-03; First posted 2020-03-05 (Actual); Last update posted 2022-07-28 (Actual); Status verified 2022-07

CONDITIONS: COPD Exacerbation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The Headstart Test system is an in vitro diagnostic test intended for self-testing for the detection of five biomarkers of infection in the urine of patients diagnosed with chronic obstructive pulmonary disease (COPD).

Patient urine testing will be conducted daily to establish a patient baseline biomarker profile and provide ongoing monitoring for changes in the biomarker profile. Headstart results will be used as an aid in monitoring and early detection of pulmonary exacerbation.

DETAILED DESCRIPTION:
Patients will be asked to collect and test a daily urine sample using a novel testing system (HeadStart Test system) in addition to answering questions abut their daily COPD symptoms for 6 months.

In summary, this study aims to validate a novel non-invasive point of care (near-patient) testing system, to allow people with COPD to detect pulmonary exacerbations by measuring urinary biomarkers. If successful, we hope that this will provide patients with an easy to use device, which will empower patients and their caregivers to treat exacerbations at an earlier stage, with potential health and economic benefits.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 40 years or over.
2. Diagnosis of COPD Stage 2-4 (GOLD I-IV) by spirometry.
3. Be a frequent exacerbator ie. ≥2 moderate exacerbations in the past 12 months.
4. Current or ex-smokers with a smoking history of at least 10 pack-years.
5. Be willing and able to comply with study procedures and be available for study visits
6. Be able to use a 'smart phone'.
7. Be able to give written consent.
8. Able to understand written and spoken English. -

Exclusion Criteria:

1. Inability to give written informed consent
2. Known respiratory disorders other than COPD which, in the opinion of the investigator, is the main contributor to patient's symptoms (e.g. asthma, lung cancer, sarcoidosis and other interstitial lung disease (ILDs), tuberculosis, lung fibrosis, cystic fibrosis, and non-COPD related bronchiectasis).
3. Known history of significant systemic and other organ-related disease, other than COPD, which in the opinion of investigator, is likely to interfere with the study or impact on subject safety (e.g. severe rheumatoid arthritis and Lupus, kidney, liver, endocrine, psychological disorders).
4. Known to be severely alpha-1-antitrypsin deficient (PI SZ or ZZ).
5. Having undergone lung surgery (e.g. lung volume reduction, lobectomy) within the last 6 months.
6. Have cancer, or other terminal condition, which, in the opinion of investigator, has a mortality of 12 months or less.
7. Have, in the opinion of the investigator, evidence of alcohol, drug or solvent abuse.
8. Taking high dose oral corticosteroid medication (equivalent to daily dose of ≥10mg of prednisolone) for more than 3 consecutive months.
9. Pregnancy
10. Participation in an interventional clinical study within 3 months of Visit 1 or participation in a study using an investigational medicinal product (IMP) either in the previous 3 months or in the interval from last using the IMP to 5 times its half-life.
11. Patients with other significant lung disease, unable to consent, unable to use the technology (e.g. inability to use the IVD device, or complete the questionnaires), or at the Clinician's discretion for other more significant medical/social reasons.

    -

Min Age: 40 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: COPD patients, Stage 2-4 (GOLD I-IV) by spirometry, with a history of exacerbations (≥2 moderate exacerbations in the past 12 months).
Sampling Method: Non-Probability Sample
Enrollment: 86 (Actual)
Dates: Start 2019-11-19 (Actual); Primary Completion 2022-02-15 (Actual); Study Completion 2022-07-24 (Actual)

PRIMARY OUTCOMES:
Headstart IVD performance | 6 months
  To determine whether the Headstart Test system can accurately diagnose an acute exacerbation of COPD prior to the onset of a clinically confirmed event. (Defined as need for antibiotics and/or Oral Corticosteroids (OCS) and/or attendance to hospital (GOLD 2019).

CONTACTS AND LOCATIONS:
Locations (1):
- Institute for Lung Health, Glenfield Hospital, Leicester, Leicestershire, United Kingdom